CLINICAL TRIAL: NCT01274650
Title: Correlation Between Wound Volume and Depth of Decubitus Ulcers And Resting Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Edwards (Other)
Responsible Party: Sponsor-Investigator, Paul Edwards, Research Coordinator, Saint Elizabeth Regional Medical Center
Organization: Saint Elizabeth Regional Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 609-040
Record Dates: First submitted 2011-01-04; First posted 2011-01-11 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Decubitis Ulcer
MeSH Terms: interventions — Calorimetry, Indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decubitis Ulcer (Other): Patients admitted to the hospital with decubitus ulcers in the ischial, sacral, or coccyx area.
  Interventions: Procedure: Indirect Calorimetry

INTERVENTIONS:
Procedure: Indirect Calorimetry — Indirect Calorimetry
  Other Names: Patients admitted to the hospital with decubitus ulcers in the ischial, sacral, or coccyx area

SUMMARY:
Patient nutritional needs vary depending on several factors including age, sex, height, weight, injury and co-morbidities. Since injury affects energy expenditure in patients, this must be taken into account when assessing nutritional requirements. Indirect calorimetry will be used to measure energy expenditure of patients with decubitus ulcers of varying degrees. The primary objective of this study is to determine the effects of wound volume on metabolic rate and compare this to predictive equations used for estimating energy requirements.

DETAILED DESCRIPTION:
Adequate nutrition is an important aspect of wound healing because it provides an anabolic environment necessary for tissue repair. Without proper nutrition support, healing can be prolonged and even inhibited. Provision of adequate energy is essential in patients with decubitus ulcers to maximize nitrogen retention and facilitate wound healing. (1,2) There are few published studies that measure energy needs in patients with decubitus ulcers. Spinal cord injured patients are one of the few populations where studies have utilized indirect calorimetry to measure energy expenditure. Individuals with spinal cord injuries are particularly at risk for developing pressure ulcers. Liu, et al. (3) measured energy expenditure in 16 individuals with quadriplegia and pressure ulcers and in 16 individuals with quadriplegia but no pressure ulcers. Measured energy expenditure was significantly higher in subjects with quadriplegia and pressure ulcers. Additionally, pressure ulcer surface area was significantly correlated with predicted resting energy expenditure. In a study of paraplegic individuals, Alexander, et al. (4) found resting metabolic rate was significantly higher in those individuals with pressure ulcers compared to those with paraplegia without pressure ulcers. Additional research is needed to confirm these findings.

To determine nutrition requirements specific to each patient, energy needs must be estimated, taking into account weight, height, age, activity level as well as the size of the wound and the patient's co-morbidities. Although indirect calorimetry is the gold standard for measuring metabolic rate, it is impractical and time consuming to use this method to determine needs of every patient. Therefore, the clinician uses predictive formulas for estimating energy needs. The most commonly cited guideline for energy requirements for healing pressure ulcers is 30-35 kcal/kg (recommendation, National Pressure Ulcer Advisory Panel).(1) The European Pressure Ulcer Advisory Panel has also recommended a minimum of 30-35 kcal/kg.(2) Several equations have been derived to predict metabolic rate based on age, height, weight, and sex. Two of these predictive equations are the Harris Benedict (5) and the Mifflin-St. Jeor. (6) These equations can be adjusted for injury factors, but it is unclear if they fully account for the size of wound in patients with decubiti.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Saint Elizabeth Regional Burn and Wound Center
* Ulcer located in the Ischial, Sacral, Coccyx

Exclusion Criteria:

* Patient Has Signs of Infection
* Patient is receiving oxandrolone treatment or anabolic hormone treatment
* Is Patients receiving intermittent tube feedings

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Does the volume of decubitus ulcers have an effect on a patient's resting energy expenditure | 1 year
  Data obtained in this study will be analyzed using methods that enable a description of the patient population and a comparison of the results against previously formulated equations for energy expenditure. Descriptive summaries will be presented for demographic and clinical background variables, study objectives, and outcome variables and safety endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Elizabeth Regional Burn and Wound Center, Lincoln, Nebraska, United States